CLINICAL TRIAL: NCT05744817
Title: Maintenance Dose of Inspiratory Muscle Strength Training to Preserve Cardiovascular Adaptations
Brief Title: Reduced Volume of Inspiratory Resistance Training
Acronym: REVIRT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Resource availability
Sponsor: University of Arizona (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 00002581
Record Dates: First submitted 2023-02-15; First posted 2023-02-27 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-06

CONDITIONS: Hypertension
Keywords: vascular endothelium; blood pressure; inspiratory resistance training; non-pharmacological
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: All participants will perform training 5 days/week for 6 weeks. Participants will then be randomly allocated at a 1:1:1 ratio to stop training (control), or to perform training 1 or 3 days/week for the next 12 weeks.
Masking Description: Due to the nature of the study groups, blinding is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): 30 breaths/day (5 sets of 6 breaths, one minute of rest between sets), 5 days/week, for 6 weeks, then no exercise for 12 weeks
- IMST 1 day/week (Experimental): 30 breaths/day (5 sets of 6 breaths, one minute of rest between sets), 5 days/week, for 6 weeks, then 30 breaths/day (5 sets of 6 breaths, one minute of rest between sets), 1 day/week, for 12 weeks.
  Interventions: Behavioral: Inspiratory muscle strength training
- IMST 3 days/week (Experimental): 30 breaths/day (5 sets of 6 breaths, one minute of rest between sets), 5 days/week, for 6 weeks, then 30 breaths/day (5 sets of 6 breaths, one minute of rest between sets), 3 days/week, for 12 weeks.
  Interventions: Behavioral: Inspiratory muscle strength training

INTERVENTIONS:
Behavioral: Inspiratory muscle strength training — 30 breaths/day against a set resistance
  Arms: IMST 1 day/week; IMST 3 days/week

SUMMARY:
This clinical research study will investigate the dose of inspiratory muscle strength training needed to maintain cardiovascular adaptations induced by a six-week loading dose.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in the US and worldwide. Although it is well-known that lifestyle changes (e.g., diet, exercise) lower blood pressure (BP) and risk for cardiovascular events, an estimated ~98% of US adults with above-normal BP do not adhere to the recommended lifestyle behaviors. Common barriers to exercise, including lethargy, low exercise self-efficacy, fear of exercise-related pain, and lack of time, make adherence to traditional exercise strategies particularly difficult. The need for novel/different forms of exercise that are i) time-efficient, ii) well-tolerated, and iii) effective has never been greater.

Inspiratory muscle strength training (IMST) is a novel, time-efficient respiratory exercise, comprising just 5 sets of 6 inspiratory efforts with 1-minute rests between sets. This training takes just 5 mins/day, 5 sessions/wk, for a total weekly training time of 25-30 minutes. Distinct from other forms of traditional aerobic or high-intensity interval-type exercise, IMST is performed on a hand-held device in sitting or standing. Participants make repeated inspiratory efforts against a resistance and generate large negative pressures that are 2-4-fold greater than those generated during rest breathing, deep breathing, or high-intensity aerobic exercise. The investigators have shown that IMST performed 5 days/wk for 6 weeks, lowers SBP 9 ± 1 mmHg on average.

It is well known that exercise-induced adaptations plateau over time, despite increases in volume and/or intensity. Accordingly, the goal of exercise is not only to improve health, but to maintain health adaptations long term. Importantly, the dose of exercise required to improve health/performance is higher than the dose required to maintain health/performance. Given that lack of time is the most often cited reason for adults failing to initiate exercise and stopping chronic exercise participation, it is essential that any potential participant 1) appreciate the relationship between time spent exercising and health improvements and 2) understand how much exercise is needed to preserve exercise-induced adaptations to ensure an unnecessary amount of time is devoted to exercise. The investigators have shown that 6 weeks of IMST can significantly lower BP and improve respiratory strength, however, the dose needed to preserve these adaptations is unknown.

This study comprises a 6-week loading dose of IMST (5 days/week; Endpoint 1), followed by 12 weeks of IMST at a reduced dose (0, 1, or 3 days/week; Endpoint 2).

ELIGIBILITY:
Inclusion Criteria:

* 50+ years of age
* systolic blood pressure between 120-169 mmHg
* stable dose of medication (three months on the same dose)
* weight stable in the prior 3 months (<3.0 kg weight change) and willing to remain weight stable throughout the study
* absence of unstable clinical disease as determined by medical history
* owns a smartphone

Exclusion Criteria:

* current smoker (including tobacco products, vaping devices, THC, etc…)
* have an uncontrolled medical condition (e.g., cancer)
* myocardial infarction or stroke within the previous 12 months
* performs regular aerobic exercise (>4 bouts/week)
* BMI ≥ 40 kg/m2
* systolic blood pressure <120 or ≥170 mmHg
* diastolic blood pressure >100 or <60 mmHg
* Cheyne-Stokes respiration
* history of perforated eardrum
* history of glaucoma or retinopathy
* history of collapsed lung
* diagnosed with asthma
* pregnant, breastfeeding, or trying to become pregnant (self-reported)
* medications that, in the opinion of the study physician, may impact the outcomes of the study (e.g., steroids)
* does not own a smartphone or is unwilling to download the required application

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-13 (Estimated); Primary Completion 2024-06-13 (Estimated); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline to endpoint 1 (6 weeks) resting systolic blood pressure | Blood pressure will be assessed at baseline and after 6 weeks of training
  Systolic blood pressure (SBP) will be measured by absolute change from baseline. SBP will be assessed in accordance with American College of Cardiology/American Heart Association guidelines. Measurements will be taken using an automated oscillometric sphygmomanometer and will be performed in triplicate over the brachial artery of the left arm after 5 minutes of quiet rest, with 1 minute of recovery between measures. SBP will be defined as the average of the 3 pressures.
Change from endpoint 1 (6 weeks) to endpoint 2 (+12 weeks) resting systolic blood pressure | Blood pressure will be assessed after 6 weeks of training and after an additional 12 weeks of training
  Systolic blood pressure (SBP) will be measured by absolute change from endpoint 1. SBP will be assessed as described in Outcome 1.
Change from baseline to endpoint 1 (6 weeks) Nitric Oxide-mediated Endothelium Dependent Dilation (EDD) | EDD will be assessed at baseline and after 6 weeks of training
  Brachial artery Flow Mediated Dilation (BA-FMD), a well-established measure of NO-mediated endothelial function, will be measured by both relative and absolute changes from baseline. BA-FMD will be determined using high-resolution ultrasonography and analyzed with a commercially available software package. An ultrasound probe will be placed 3-6 cm proximal to the antecubital crease on the right arm and a baseline image of the right brachial artery will be obtained. Following baseline, reactive hyperemia will be produced by inflating a rapid-inflating blood pressure cuff. Brachial artery diameter change will be measured for 2 minutes following 5-min of forearm blood flow occlusion.
Change from endpoint 1 (6 weeks) to endpoint 2 (+12 weeks) Nitric Oxide-mediated Endothelium Dependent Dilation (EDD) | EDD will be assessed after 6 weeks of training and after an additional 12 weeks of training
  EDD will be assessed as described in Outcome 3

SECONDARY OUTCOMES:
Change from baseline to endpoint 1 (6 weeks) cerebrovascular reactivity (CVR) | CVR will be assessed at baseline and after 6 weeks of training
  CVR will be assessed via changes in middle cerebral artery (MCA) blood velocitywill be assessed in a reclined sitting position while breathing room air and again after 4 min of breathing a medical gas mixture with 5 % CO2 l to elicit vasodilation. A transcranial Doppler probe will be placed over the subject's temple to obtain a velocity tracing from the middle cerebral artery. After a tracing of MCA velocity is obtained and baseline measurements are recorded (while breathing room air), the subject will then switch over to breathing 5% CO2 for
Change from endpoint 1 (6 weeks) to endpoint 2 (+12 weeks) | CVR will be assessed after 6 weeks of training and after an additional 12 weeks of training
  CVR will be assessed as described in Outcome 5

CONTACTS AND LOCATIONS:
Overall Officials: Dallin Tavoian, PhD, Principal Investigator — University of Arizona
Locations (1):
- Arizona Respiratory and Neurophysiology Laboratory, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No